CLINICAL TRIAL: NCT04296916
Title: Effect of Medically Lowering Intraocular Pressure in Glaucoma Suspects With High Myopia: A Randomized Controlled Trial
Brief Title: Effect of Lowering IOP in Glaucoma Suspects With HM
Acronym: GSHM
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Xiulan Zhang, Director of Clinical Research Center, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2020KYPJ026
Record Dates: First submitted 2020-03-03; First posted 2020-03-05 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Glaucoma, Suspect; High Myopia
Keywords: Glaucoma, Suspect; High myopia; Intraocular Pressure
MeSH Terms: conditions — Ocular Hypertension

STUDY DESIGN:
Intervention Model Description: Open-label, single-center, randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Participants and physicians are not masked as to the treatment assignment. The study outcomes will be obtained by masked ophthalmic technicians according to standard protocols and read by masked graders at the End Point Adjudication Committee. The masking status of the technicians collecting data will be recorded at each study visit. The study data will be analyzed by masked researchers.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): medical reduction of IOP by eyedrops
  Interventions: Drug: IOP lowering eye drops
- control arm (No Intervention): follow up without medication

INTERVENTIONS:
Drug: IOP lowering eye drops — 1. Latanoprost 0.005% eye drops will be the first choice. If an IOP reduction of 20% is not achieved within three months, timolol 0.5% will be added as second medication. If an IOP reduction of 20% is then not achieved, alphagan 0.2% or alphagan-P 0.15% will be added. If an IOP reduction of 20% is then not achieved, the individual will be excluded from the study.
  2. If necessary, latanoprost will be switched to other prostaglandin eye drops, alphagan (or alphagan-P) will be switched to brinzolamide 1% eye drops.
  3. If necessary, latanoprost and timolol will be switched to Xalacom eye drops, timolol and alphagan will be switched to Combigan eye drops, timolol and brinzolamide will be switched to Azarga eye drops.
  4. Once daily in the evening for prostaglandin eye drops, and twice daily for other eye drops.
  Arms: Intervention arm

SUMMARY:
Currently, whether and when intraocular pressure (IOP) lowering medication should be used in glaucoma suspects with high myopia (HM) is still a dilemma. Randomized trials are required to evaluate whether IOP lowering influences the incidence of glaucoma suspect progression in HM eyes.

DETAILED DESCRIPTION:
HM is associated with increased prevalence of glaucoma. However, accurate diagnosis of glaucoma in HM is a challenge. More and more viewpoints had been raised that HM eyes with optic disc head damage or/and visual field (VF) defects should been classified as glaucoma suspects.

IOP is the only modifiable parameter in glaucoma and glaucoma suspect patients. However, the decision to begin treatment to lower IOP in the glaucoma suspect patient is complex, especially for glaucoma suspects with HM. There are lack of guideline and consensus of treatment choices. Therefore, it is necessary to investigate the effect of medically IOP lowering on the progression of glaucoma suspects with HM.

ELIGIBILITY:
Inclusion Criteria:

1. Aged between 35 and 65 years.
2. Diagnosed with high myopia (spherical equivalent ≤ -8.00 diopters or axial length ≥ 26.5 mm).
3. Diagnosed with glaucoma suspect, which cannot be explained by myopic macular changes, or other retinal and neurologic condition.
4. IOP ≥ 12 mmHg and ≤ 24mmHg on at least 2 visits, as measured by Goldmann applanation tonometry.
5. An open anterior chamber angle as based upon gonioscopy.
6. Best corrected visual acuity (BCVA) ≥ 6/12.

Exclusion Criteria:

1. Allergy to prostaglandins.
2. Advanced VF loss (MD worse than 16 dB) or a threat to fixation (sensitivity 10 dB or worse affecting either or both test points closest to the point of fixation in the upper hemifield and at either or both of the corresponding test points in the lower hemifield) in either eye.
3. Previous IOP-lowering surgery in the study eye (i.e. trabeculectomy, Ahmed glaucoma valve implantation, any laser trabeculoplasty).
4. Previous cataract surgery in the study eye.
5. Previous corneal refractive surgery in the study eye.
6. Clinically significant or progressive retinal disease such as proliferative diabetic retinopathy, retinal detachment, central retinal vein occlusion, or retinitis pigmentosa in the study eye.
7. Chronic, recurrent or severe inflammatory eye disease in the study eye (from screening), such as chronic or recurrent uveitis.
8. Obvious corneal and iris lesions, or severe cataracts interfering with fundus examinations, or monophtalmia.
9. Need for ocular surgery/laser or anticipated need for cataract surgery that would influence the ophthalmological parameters measured in this study during the study period.
10. Other serious systemic diseases (i.e. hypertension, heart disease, diabetes, or rheumatic immune system diseases).
11. Pregnant or nursing women.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2020-04-17 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
The number of subjects whose visual filed progressed during the follow up | 36 months

SECONDARY OUTCOMES:
The number of subjects whose optic nerve head morphology including the retinal nerve fiber layer (RNFL) and ganglion cell-inner plexiform layer (GCIPL) changed during the follow up | 36 months
The number of subjects whose myopic maculopathy progressed during the follow up | 36 months
The number of subjects whose visual function and quality of life changed during follow up | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Xiulan Zhang, MD, PhD, Principal Investigator — Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Leske MC, Hyman L, Hussein M, Heijl A, Bengtsson B. Comparison of glaucomatous progression between untreated patients with normal-tension glaucoma and patients with therapeutically reduced intraocular pressures. The effectiveness of intraocular pressure reduction in the treatment of normal-tension glaucoma. Am J Ophthalmol. 1999 May;127(5):625-6. No abstract available. PMID 10334369
- [Result] Garway-Heath DF, Crabb DP, Bunce C, Lascaratos G, Amalfitano F, Anand N, Azuara-Blanco A, Bourne RR, Broadway DC, Cunliffe IA, Diamond JP, Fraser SG, Ho TA, Martin KR, McNaught AI, Negi A, Patel K, Russell RA, Shah A, Spry PG, Suzuki K, White ET, Wormald RP, Xing W, Zeyen TG. Latanoprost for open-angle glaucoma (UKGTS): a randomised, multicentre, placebo-controlled trial. Lancet. 2015 Apr 4;385(9975):1295-304. doi: 10.1016/S0140-6736(14)62111-5. Epub 2014 Dec 19. PMID 25533656
- [Result] Leske MC, Heijl A, Hyman L, Bengtsson B. Early Manifest Glaucoma Trial: design and baseline data. Ophthalmology. 1999 Nov;106(11):2144-53. doi: 10.1016/s0161-6420(99)90497-9. PMID 10571351
- [Derived] Lin FB, Da Chen S, Song YH, Wang W, Jin L, Liu BQ, Liu YH, Chen ML, Gao K, Friedman DS, Jonas JB, Aung T, Lv L, Liu YZ, Zhang XL; GSHM study group. Effect of medically lowering intraocular pressure in glaucoma suspects with high myopia (GSHM study): study protocol for a randomized controlled trial. Trials. 2020 Sep 29;21(1):813. doi: 10.1186/s13063-020-04748-7. PMID 32993769